CLINICAL TRIAL: NCT05798143
Title: Developing Translational Biomarkers to Predict Clinical Response in Treatment-resistant Depression: Towards a Personalized, Plasticity-enhancing Accelerated Neuromodulation
Brief Title: Translational Biomarkers in Accelerated Neuromodulation for Treatment-resistant Depression
Acronym: ReModula
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ITAB - Institute for Advanced Biomedical Technologies (Other)
Responsible Party: Principal Investigator, Mauro Pettorruso, Dr, ITAB - Institute for Advanced Biomedical Technologies
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: remodula
Record Dates: First submitted 2023-03-03; First posted 2023-04-04 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: Treatment Resistant Depression
Keywords: Treatment resistant depression; accelerated repetitive transcranial magnetic stimulation; arTMS; TRD; biomarkers; neuroplasticity
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Active arTMS treatment (Experimental): rTMS is a non-invasive brain stimulation technique. It will be used a MagPro R30 with the Cool-B-70 figure-of-eight coil (MagVenture, Falun, Denmark).
  Interventions: Device: Accelerated Repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Accelerated Repetitive Transcranial Magnetic Stimulation — rTMS is a non-invasive brain stimulation technique. It will be used a MagPro R30 with the Cool-B-70 figure-of-eight coil (MagVenture, Falun, Denmark).
  Other Names: arTMS

SUMMARY:
Background: 30-50% of patients with Major Depressive Disorder (MDD) do not respond adequately despite two or more antidepressant treatments with proper dosage and timing of administration, configuring a condition of Treatment-Resistant Depression (TRD). Repetitive Transcranial Magnetic Stimulation (rTMS) is a neuromodulation technique that uses a magnetic field to stimulate focal cortical brain regions and it has been approved by the FDA for the treatment of TRD. Accelerated rTMS (arTMS) protocols involve multiple daily sessions of rTMS and they have been shown to be equally effective and safe compared to rTMS protocols, with reduced administration time and potentially faster antidepressant efficacy.

Objectives: The main aim of this study is to identify MDD endophenotypes/biotypes predictive of response to accelerated treatment of rTMS to better characterize the clinical correlates of response in patients with TRD.

Eligibility: Subjects between 18 and 65 years suffering from TRD in stable psychopharmacological treatment for at least one month.

Design: This clinical trial includes three phases: 1) a screening phase; a rTMS continued treatment phase; and a follow-up.

In order to be enrolled, participants will be screened with:

* Medical history to assess the existence of the inclusion criteria and exclude any medical conditions that could contraindicate treatment with arTMS
* Questionnaires

After being enrolled, baseline data will be collected. In particular, participants will be administered:

* Questionnaires
* Functional MRI
* Cognitive tasks
* Eye examination with Electroretinography (ERG)
* Blood sampling
* Salivary cortisol sampling

Repetitive TMS will be delivered during 5 outpatient treatment days (4 times/die).

After treatment patients will be contacted by telephone on a weekly basis for the first 3 weeks, to carry out an assessment of the clinical condition.

A follow-up visit, in the clinic, will be carried out after 21 days from the last stimulation (Friday), with the administration of psychometric scales.

Blood samples will be taken on the first day of stimulation and the day after the last stimulation.

Salivary cortisol sampling will be taken before the start of the stimulation protocol, after the first stimulation day and immediately after the last stimulation session foreseen by the protocol.

fMRI will be performed during baseline and at the end of treatment. ERG will be performed before the start of the stimulation protocol, after the first stimulation and immediately after the last stimulation session foreseen by the protocol. Patients will undergo ERG again during the follow-up visit at 21 days.

Treatment includes:

* rTMS: A brief electrical current passes through the coil placed on the head. At each day, participants will receive four rTMS sessions (36 min), with a 55 min interval between sessions.
* MRIs: Patients will undergo two MRI sessions lasting 45 min. Blood pressure and respiratory rate will be recorded before the examination. During fMRI, patients will be asked to perform tasks.
* Eye examination with Electroretinography (ERG)
* Blood and salivary sampling.
* Screening tests and questionnaires.

DETAILED DESCRIPTION:
The main aim of the study is to identify MDD endophenotypes/biotypes predictive of response to accelerated treatment of rTMS to consolidate the use of a cost-effective protocol and to better characterize the clinical correlates of response in patients with TRD. In addition, the present study proposes the following secondary objectives: A) identification of applicable and reliable peripheral biomarkers related to endophenotypes/biotypes, exportable in clinical practice to predict response to treatment; B) evaluation of potential synergistic, additive or antagonistic effects of MDD pharmacotherapies when used in combination with neuromodulation interventions.The study includes 3 psychiatric assessments with psychometric testing: T0 (enrollment), T1 (day 6), T2 (week 3, follow-up). At T0 (enrollment) the Researcher will fully inform the patient about the study, obtaining the patient's informed consent to participate in the study, and will determine the patient's eligibility. Patients will also undergo a battery of cognitive tasks aimed at measuring any changes caused by the neuromodulatory action of arTMS. During T1 (day 6), and T2 (3 weeks) the patient will again undergo the tests and neurocognitive evaluations. arTMS protocol involves 20 rTMS sessions (4/daily for 5 consecutive days, each session lasts 35 min with an interval of 55 min). Coil is placed on the left dorsolateral prefrontal cortex (LDLPFC), trains have a frequency of 10 Hz and a intensity of 120% of the individual resting motor threshold.

To investigate the possible effects of arTMS on brain connectivity, patients will undergo a functional neuroimaging study based on fMRI on T0 and T1. MDD biomarkers measurable by ERG could represent a valid aid in the personalization of treatments. ERG will be performed before the start of the stimulation protocol (T0), after the first stimulation and immediately after the last stimulation session foreseen by the protocol. Patients will undergo ERG again during the follow-up visit at 21 days (T2). Blood samples will be taken on the first day of stimulation (T0) and the day after the last stimulation to identify reliable peripheral biomarkers related to endophenotypes/biotypes, exportable in clinical practice to predict response to treatment. Salivary cortisol sampling will be taken before the start of the stimulation protocol (T0), after the first stimulation day and immediately after the last stimulation session foreseen by the protocol. Some variations in neuroendocrine biomarkers such as cortisol seem to be predictive of response to arTMS treatment. The analysis of the neuroimaging, ERG and peripheral data will lead to identify MDD endophenotypes/biotypes predictive of response to accelerated treatment of arTMS.

ELIGIBILITY:
Inclusion Criteria:

* Current diagnosis of Major Depressive Disorder (MDD), based on the Diagnostic and Statistical Manual of Mental Disorder - Fifth Edition (DSM-5);
* Subjects without clinical response to at least two antidepressant treatments administered at adequate dosage and duration during the current episode;
* Stable psychopharmacological treatment for at least one month.

Exclusion Criteria:

* Co-morbidity with organic diseases that could interfere with magnetic stimulation safety (epilepsy, brain lesions or diseases, previous neurosurgery, metal grafts, cardiac devices) based on applied procedure guidelines;
* Diagnosis of Substance or Alcohol Use Disorder (DSM-5) in the past 6 months;
* Substances of abuse or alcohol acute intoxication or abstinence;
* Co-morbidity with significant organic or neurological diseases;
* Personal or familiar (1st degree relatives) medical history of seizures;
* Significant eye diseases that could interfere with ERG execution;
* For female patients: Pregnancy/breastfeeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-02-28 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in psychometric test indicator of depression - MADRS | Baseline; each 1 day of treatment ; at 1, 2, 3 and 4 weeks.
  Montgomery Asberg Depression rating scale (MADRS - 10 items - score 0-60) to measure relevance of mood, concentration, physical and sleep symptoms
Changes in psychometric test indicator of depression - HAM-D 21 | Baseline; 1 week; 4 weeks
  Hamilton Depression Scale (HAM-D - 21 items - score 0-69) to assess relevance and pervasiveness of depressive symptoms
Changes in neuroplasticity - structural RM and fMRI (physiological parameter) | Baseline; day 6
  Functional MRI (which requires a preliminary structural MRI) produces images of the brain both in a "resting state" and when it is engaged in producing movements, sensations or when concentrated in activities involving emotional and cognitive responses. It is based on the ability to capture the signals emitted by hydrogen atoms when they are subjected to a magnetic field.
Changes in neuroplasticity - DTI (physiological parameter) | Baseline; day 6
  Diffusion Tensor Imaging (DTI) techniques to assess the integrity of white matter tracts between brain regions. DTI data, accompanied by fMRI studies, in subjects with MDD are indicative of reduced functional connectivity between cortical and subcortical structures.
  It is based on the principle of Brownian motion of water molecules, the signal is directly proportional to the integrity of the myelin sheath.
Changes in responsivity of nervous tissue (physiological parameter) | Baseline; 4 weeks
  ERG will be performed to gain an easy access to structural and functional nervous tissue alterations, usually observed in MDD patients and partially reversible with antidepressant treatment. The ERGs records the electrical activity following single light stimuli (flash), able to provide an indication of the activity of the external (cones, rods) and intermediate (amacrine, bipolar cells) layers of the retina
Rate of genetic polymorphism predictor of treatment response | Baseline; day 6
  Genetic tests investigating polymorphism (5-HT2A, 5-HT1A and BDNF receptors), possible predictors of antidepressant treatment response
Change in BDNF level (physiological parameter) | Baseline; day 6
  BDNF levels will be evaluated by collecting a venous blood sample. BDNF is a member of the nerve growth factor (NGF) family of neurotrophic growth factors. Low levels of peripheral BDNF and NGF have been reported in mood disorders and other psychopathological conditions with normalization after antidepressant treatment or mood stabilization. The increase in serum levels of BDNF seems to reflect the concomitant activation of BDNF synthesis that accompanies the neuronal remodeling triggered by the suspension of alcohol intake and suggests that the synthesis of BDNF may have a role in the long-term maintenance of alcohol abstention. BDNF measurements will be calculated in pg/ml
Change in pro-BDNF (physiological parameter) | Baseline; day 6
  Pro-BDNF is the precursor of BDNF and it acts as a repository of mature BDNF and acts itself by inducing neuronal thinning. Pro-BDNF levels will be evaluated by collecting a venous blood sample. Pro-BDNF measurements will be calculated in ng/ml.
Changes in peripheral biomarkers - HPA axis (blood) | Baseline; day 6
  Hypothalamic-Pituitary-Adrenal axis will be evaluated assessing blood cortisol (mcg/dL) and ACTH (mcg/dL) levels
Changes in peripheral biomarkers - HPT axis (FT3/FT4) | Baseline; day 6
  Hypothalamic-Pituitary-Thyroid aill be evaluated assessing, FT3 (pmol/L) and FT4 ( pmol/L) levels
Changes in peripheral biomarkers - HPT axis (TSH) | Baseline; day 6
  Hypothalamic-Pituitary-Thyroid aill be evaluated assessing TSH (μIU/mL)
Changes in peripheral biomarkers - HPA axis (saliva) | Baseline; day 6
  Hypothalamic-Pituitary-Adrenal axis will be evaluated assessing salivary (µL) levels of cortisol
Changes in peripheral biomarkers - C reactive protein (physiological parameter) | Baseline; day 6
  C reactive protein, that indicates the inflammation degree, in mesured in mg/L.

SECONDARY OUTCOMES:
Cognitive Performance Using the THINC-it Tool | Baseline, 4 weeks
  THINC-it (an acronym), include nclude the Spotter task (Choice Reaction Time), Symbol Check task(1-back test),Trails task(Trails Making Test B), and Codebreaker task (Digit Symbol Substitution Test).Z-value indicates the performance result (higher z higher performance)
Trait scales - TEMPS-A-brief Italian Version | Baseline
  Temperament Evaluation of Memphis, Pisa and San Diego Autoquestionnaire brief version (TEMPS-A-brief Italian Version - subscales' score: cyclothymic 0-12; depressive 0-8; irritable 0-8; hyperthymic: 0-8; anxious 0-3): a 39 items scale to investigate temperamental traits
Trait scales - BIS-11 | Baseline
  Barratt Impulsiveness Scale, Version 11 (BIS-11, 30 item - score 30-120) to evaluate temperamental impulsive traits. BIS-11 consists in 3 subscale: "Attentional Impulsivity", "Motor Impulsivity" and "Nonplanning Impulsivity"
Trait scales - CTQ-28 items | Baseline
  Childhood Trauma Questionnaire (CTQ-28 items - score 0-112) to evaluate childhood and adolescence abuses and trauma
Trait scales - TAS-20 | Baseline
  Toronto Alexithymia Scale (TAS-20 - 20 items - score 20-100) to assess emotional self-awareness
Trait scales - BFQ-R | Baseline
  Big Five Questionnaire (BFQ-R 60 items - score 60-300) to assess the big five personality traits (extraversion, agreeableness, conscientiousness, neuroticism, and openness)
State scales - ASMR | Day 1,2,3,4,5
  Altman Self-Rating Mania Scale (ASRM - 5 item - score 0-20) to evaluate presence and relevance of manic symptoms
State scales - TMS collateral effect scale | After each TMS session
  TMS collateral effect scale, to evaluate possible collaterality due to magnetic stimulation
State scales - YMRS | Baseline; 1 week; 4 weeks
  Young Mania Rating Scale (YMRS - 11 item - score 0-44) investigating symptoms of mania
State scales - BPRS | Baseline; 1 week; 4 weeks
  Brief Psychiatric Rating Scale (BPRS - 24 items - score 24-168) for a global psychopathological assessment
State scales - SHAPS | Baseline; 1 week; 4 weeks
  Snaith-Hamilton Pleasure Scale (SHAPS - 14 items - score 0-42) to estimate hedonic tone
State scales - BHS | Baseline; 1 week; 4 weeks
  Beck Hopelessness Scale (BHS- 20 items - score 0-20) to evaluate negative attitudes towards the future and pessimism
State scales - ISI | Baseline; 1 week; 4 weeks
  Insomnia Severity Index (ISI - 5 items - score 0-28) to assess quality of sleep
State scales - SDS | Baseline; 1 week; 4 weeks
  Sheehan Disability Scale (SDS 5 items - score 0-30) to measure disability perceived by patient
State scales - CGI-S | Baseline; 1 week; 4 weeks
  Clinical Global Impression - Severity scale (CGI-S - score 1-7) to estimate clinical disease entity
State scales - LAPS | Baseline; 1 week; 4 weeks
  Leuven affect and pleasure scale (LAPS 16 items - score 0-160) to assess positive and negative affective and hedonic tone
State scales - SF | Baseline; 1 week; 4 weeks
  Health Questionnaire (SF-12 items - score 12-47) to evaluate quality of life
Changes in psychometric test indicator of depression - HAM-A 21 | Baseline; 1 week; 4 weeks
  Hamilton Anxiety Scale (HAM-A - 21 items) to assess anxiety relevance

CONTACTS AND LOCATIONS:
Locations (1):
- ITAB, Chieti, Italy

IPD SHARING:
Plan to Share IPD: No